CLINICAL TRIAL: NCT03445585
Title: A Resource of Blood and Other Biospecimens of Patients With Cholestatic Liver Disease and Unaffected Individuals
Brief Title: Biobank for Cholestatic Liver Diseases.
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Konstantinos N. Lazaridis, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 16-005892
Record Dates: First submitted 2017-02-14; First posted 2018-02-26 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Primary Sclerosing Cholangitis; Primary Biliary Cirrhosis; Cholangiocarcinoma; Liver Cancer
MeSH Terms: conditions — Cholangitis, Sclerosing; Liver Cirrhosis, Biliary; Cholangiocarcinoma; Liver Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — This study will collect bile and bile duct cells during ERCP procedures, residual liver tissue from liver transplants, blood, stool, and urine.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (4):
- Primary Sclerosing Cholangitis: Patients with a diagnosis of primary sclerosing cholangitis (PSC).
- Primary Biliary Cirrhosis/Cholangitis: Patients with a diagnosis of primary biliary cirrhosis (PBC).
- Control group 1: Patients who do not have PBC or PSC but do have another form of chronic liver disease.
- Control group 2: Patients without liver disease.

SUMMARY:
This study is a biobank of specimens and clinical data for use in current and future research to better understand the cholestatic liver diseases primary biliary cirrhosis/cholangitis (PBC) and primary sclerosing cholangitis (PSC).

DETAILED DESCRIPTION:
This study is a biobank of specimens and clinical data for use in current and future research to better understand the cholestatic liver diseases primary biliary cirrhosis/cholangitis (PBC) and primary sclerosing cholangitis (PSC).

Blood, saliva, stool, and urine samples will be collected periodically during patient visits or via a mail-home kit. Bile and bile duct cells will be collected during clinically necessary Endoscopic Retrograde Cholangiopancreatography (ERCP) procedures. Anticipated research will focus on multi-omics assessments of biospecimens to better define how these diseases start and progress in order to develop novel tests for early detection of complication and better disease prognostication.

ELIGIBILITY:
Inclusion Criteria:

PSC

* Patients diagnosed with PSC and who are between the age of 18 and 85 at time of enrollment in the study.
* The diagnosis of PSC will be based on standard PSC criteria including clinical and biochemical evidence of chronic cholestasis of at least six months duration, positive cholangiographic findings, and compatible liver biopsies if available.
* Patients with PSC who have undergone orthotopic liver transplantation will be offered enrollment except for collection of bile - please see below under Exclusion Criteria.
* Women with PSC of childbearing potential and pregnant women will be offered enrollment because there is no risk to an unborn child in this investigation.

PBC

* Patients diagnosed with PBC and who are between the age of 18 and 85 at time of enrollment in the study.
* The diagnosis of PBC will be based on standard PBC criteria including clinical and biochemical evidence of chronic cholestasis of at least six month duration, positive anti-mitochondrial antibodies in serum and compatible liver biopsies, if available.
* Patients with PBC who have undergone orthotopic liver transplantation will be offered enrollment except for collection of bile - please see below under Exclusion Criteria.
* Women with PBC of childbearing potential and pregnant women will be offered enrollment because there is no risk to an unborn child in this investigation.

Controls

* Controls without history of PBC, PSC, or evidence of other chronic liver disease of either gender that participate in this study will be between the ages of 18 and 85.

Liver Disease Controls

* Patients without history of PBC or PSC but do have evidence of other chronic liver disease of either gender will be offered participation in this study if between the ages of 18 and 85.

Exclusion Criteria (all subjects):

* PBC or PSC patients with known and overlapping other chronic liver diseases
* Patients unable to provide informed consent
* Prisoners and institutionalized individuals

Exclusion Criteria (for bile collection during ERCP)

* PSC with orthotopic liver transplantation
* History of Roux en Y

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with PBC, PSC, controls without liver disease, and with other chronic liver disease without history of PBC or PSC seen or followed at Mayo Clinic will be invited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 9150 (Estimated)
Dates: Start 2017-01; Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants in the study. | 20 years
  Number of participants in the study.

SECONDARY OUTCOMES:
Number of samples collected (per type). | 20 years
  Number of samples collected (blood, urine, stool, bile, bile duct cells)
Number of clinical phenotypes and/or endpoints observed (per category) | 20 years
  Number of clinical phenotypes and/or endpoints observed (i.e. disease progression, liver cancer development)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Lazaridis, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No